CLINICAL TRIAL: NCT05829486
Title: The Effects of Ketamine and Propofol and Remifentanil and Propofol Combinations on Integrated Pulmonary Index During Sedation in Gastroscopy
Brief Title: Integrated Pulmonary Index in Gastroscopic Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Zuhal Çavuş, Medical doctor, principal investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 147/22
Record Dates: First submitted 2023-03-31; First posted 2023-04-25 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Endoscopy
Keywords: sedation; respiratory complications; ambulatory anesthesia
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ketaprop: At the beginning of anesthesia, 0.25 mg/kg ketamine and 0.75 mg/kg propofol will be administered.
  Interventions: Procedure: gastroscopy
- remiprop: At the beginning of anesthesia, 1 mcg/kg of remifentanil and 0.75 mg/kg propofol will be administered.
  Interventions: Procedure: gastroscopy

INTERVENTIONS:
Procedure: gastroscopy — anaesthetic management of ambulatory endoscopic procedures

SUMMARY:
Various complications are the leading cause of morbidity in sedation practices in endoscopic procedures, and guidelines recommend continuous monitoring of circulation, respiratory function, and ventilation. Integrated Pulmonary Index (IPI), one of the methods that can be used in this monitoring, gives a single numerical value obtained by continuous and simultaneous joint mathematical analysis of Oxygen saturation, End-tidal carbon dioxide concentration, respiratory rate, and heart rate values and is a good monitorization in these interventions. and provides tracking. In this study, the aim is to determine the role of IPI in the diagnosis and follow-up of respiratory complications in patients who were sedated during gastroscopy procedures.

DETAILED DESCRIPTION:
IPI EtCO2 is a monitoring method consisting of respiratory rate, SPO2 and heart rate parameters. While EtCO2 is measured with nasal capnography, SPO2, heart rate, respiratory rate are measured with finger probe and it will show instant measurement of respiratory status. IPI takes values between 1-10. An IPI value of 8 and above will indicate normal values, a value between 5-7 will indicate that the respiratory status of the patient should be carefully examined and intervened if necessary, values of 4 and below will definitely indicate that the patient's respiratory status should be intervened.

Blood pressure measurement will be made with a sphingmomanometer noninvasively at certain time intervals with the help of a cuff that will be placed on the patient's arm area.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3 risk scored patients,
* patients over the age of 18 who will undergo endoscopic intervention

Exclusion Criteria:

* Patients who need mechanical ventilator support,
* patients who need emergency endoscopic intervention,
* patients with a history of substance abuse,
* patients with a history of allergy to the drugs to be used,
* pregnant women will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: over the age of 18 who will undergo endoscopic intervention
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
respiratory complications comparing different sedative groups | Measurements will be in 4 time frames; before induction anesthesia, 5 minutes after the induction of sedation, 10 minutes after the induction, 5 minutes after the end of the procedure
  Comparison of sedation safety and efficacy of Ketamine and Propofol and Remifentanil and Propofol administration to be applied to patients in endoscopy by using integrated pulmonary index (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: zuhal çavuş, MD, Principal Investigator — gaziosmanpasa TREH; döndü genç moralar, MD, Study Director — gaziosmanpasa TREH
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided